CLINICAL TRIAL: NCT05438667
Title: A Prospective, One Arm Clinical Study on the Safety, Efficacy and Pharmacokinetics of KRAS Mutant Antigen Specific TCR-T Cells in the Treatment of Advanced Solid Tumors.
Brief Title: TCR-T Cell Therapy on Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2022]01-01
Record Dates: First submitted 2022-06-07; First posted 2022-06-30 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; PK/PD; TCR-T; Safety; efficacy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T treatment group (Experimental): Within 3-5 days after pretreatment, subjects will receive a single TCR-T infusion with an infusion dose of about 1 × 10⁹～1 × 10¹⁰.Once every 12 hours within 24 hours after TCR-T cell infusion, recombinant human interleukin-2 will be injected intravenously for 5 days. After 3 months of treatment, the patient's condition was evaluated. If the subject did not occur tumor progression and did not occur adverse events (AEs) of level 3 or higher, a second TCR-T cell reinfusion can be performed .
  Interventions: Biological: TCR-T therapy

INTERVENTIONS:
Biological: TCR-T therapy — 1.Preprocessing strategy：
  1. Cyclophosphamide: 300-450mg/m², dissolved in 100ml 0.9% sodium chloride saline, intravenous drip for 60minutes, and 0.4g Mesna injected at 0hour, 4hours and 8 hours after cyclophosphamide,4days and 5 days before TCR-T cell infusion.
  2. Fludarabine: 30mg/m² , dissolved in 100ml 0.9% sodium chloride saline, intravenous drip for 30minutes before 3 to 5days before TCR-T cell infusion.
  2.Within 3-5 days after pretreatment, subjects will receive a single TCR-T reinfusion with an infusion dose of about 1 × 10⁹～1 × 10¹⁰.
  3.Once every 12 hours within 24 hours after TCR-T cell infusion, recombinant human interleukin-2 (injection unit: 500000 units /m², once every 12 hours, subcutaneous injection) will be injected intravenously for 5 days (10 times in total).
  4.After 3 months of treatment, If the subject did not occur tumor progression and did not occur adverse events (AEs) of level 3 or higher, a second TCR-T cell reinfusion can be performed.

SUMMARY:
The primary aim of this study is to evaluate the efficacy of KRAS mutant antigen specific TCR-T cells in the treatment of patients with advanced solid tumors.

The secondary aim is to evaluate the pharmacokinetic/pharmacodynamic characteristics of TCR-T cell therapy in patients with advanced solid tumors and the survival of TCR-T cells.

The investigators will evaluate the changes of tumor microenvironment after treatment of advanced solid tumors with KRAS mutant antigen specific TCR-T cells; Evaluating the correlation between cytokines and the occurrence of CRS and neurotoxicity

DETAILED DESCRIPTION:
1.This study is a prospective and single arm clinical study. In this trial, 18 patients with advanced solid tumors with KRAS G12V or G12D mutations and matching HLA-A subtypes are recruited for autologous Tumor-T Cell Receptor (TCR) -Mediated T Cells therapy(TCR-T) therapy.Within 3 - 5 days after pretreatment, subjects will receive a single TCR-T infusion with an infusion dose of about 1 × 10⁹～1 × 10¹⁰. Once every 12 hours within 24 hours after TCR-T cell infusion, recombinant human interleukin-2 will be injected intravenously for 5 days .

After 3 months of treatment, the patient's condition was evaluated. If the subject did not occur tumor progression and did not occur adverse events (AEs) of level 3 or higher, a second TCR-T cell reinfusion can be performed based on researcher's judgment (informed consent form needs to be signed again).

The study will evaluate the safety of TCR-T treatment by observing adverse events after cell therapy; evaluate the effectiveness of TCR-T compared to the results or historical data of the subject's own previous standard treatment regimen;and collect blood before and after cell infusion, measure the number and activity of TCR-T cells, and evaluate the pharmacokinetic (PK) characteristics of TCR-T.

ELIGIBILITY:
Inclusion Criteria：

1. Age greater than 18 years old；
2. Subjects with advanced solid tumors confirmed by histology/cytology who have failed standard treatment, are intolerant to standard treatment, or for whom no standard treatment exists. . Non-small cell lung cancer: Recurrent/metastatic non-small cell lung cancer previously treated with platinum-based chemotherapy and/or immunotherapy and/or anti-angiogenic therapy; ii. Pancreatic cancer: Recurrent/metastatic pancreatic cancer that has failed at least one prior systemic therapy; iii. Colorectal cancer: Recurrent/metastatic colorectal cancer that has failed at least two prior systemic therapies (including oxaliplatin, irinotecan, fluoropyrimidine-based agents, anti-angiogenic drugs, etc.); iiii. Other tumors: Other advanced solid tumors that have failed standard treatment, are intolerant to standard treatment, or for which no standard treatment exists;
3. Previous tissue pathology or peripheral blood testing confirmed the presence of KRAS G12V or G12D mutations with matching HLA subtypes；
4. Expected survival duration of more than 3 months；
5. Eastern Cooperative Oncology Group( ECOG )score ≤2；
6. All participants voluntarily participate in this study and sign an informed consent. And the subjects have good compliance and can cooperate with investigators follow-up study.
7. Patients at least have had at least one measurable lesion as defined by RECIST v1.1 criteria；
8. Female participants can not be pregnant or lactating and their serum or urine human chorionic gonadotropin tests must be negative within 72 hours prior to study enrollment；All subjects must be using a medically accepted means of contraception ( (e.g., oral contraceptives, intrauterine device) during the course of this study and for at least 3 months after completion of study therapy.
9. Organ function and bone marrow reserve are in good condition, and the following requirements must be met:

1)Absolute neutrophil count≥1.5×10⁹/L, Absolute lymphocyte count ≥0.5×10⁹/L；2)Platelet count≥50×10⁹/L；3)Hemoglobin≥90g/L；4)Bilirubin < 1.5 times upper limit of normal（Bile duct obstruction due to tumor compression were excluded)；5)Serum creatinine ≤ 1.5 times the upper limit of normal range or creatinine clearance ≥ 60 mL/min.6)Serum alanine aminotransferase or aspartate aminotransferase is < 2.5 times the upper limit of the normal value (ULN) (if patients with liver metastasis, ≤5 times the ULN).7)Coagulation function normalised：INR≤1.5，PTT<1.2 times the upper limit of normal（Tumor - related anticoagulant therapy was excluded).

Exclusion Criteria:

1. Intracranial metastasis or Patients with moderate or severe hydrothorax need drain placement to relieve symptoms.
2. Active pulmonary tuberculosis
3. Human immunodeficiency virus (HIV) positive；
4. Active Hepatitis B or Hepatitis C infection；
5. Pregnant women and lactating females；
6. Previous or concurrent history of other malignant tumors. Exceptions include curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy;
7. Patients with central nervous metastases；
8. Serious, uncontrolled comorbidities that may affect protocol compliance or interfere with interpretation of results，or any serious medical condition that may affect the safety of the subjects ;
9. History of clinically significant respiratory diseases or other respiratory diseases that seriously affect Pulmonary function;
10. Any active autoimmune disease,any condition requiring steroid hormones or immunosuppressive therapy( including but not limited to systemic lupus erythematosus, sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc., require > 10 mg/D of prednisone or equivalent hormone）
11. A history of organ transplantation；
12. A history of myocardial infarction and severe arrhythmia within six months；Ineligible also includes uncontrolled hypertension, coronary heart disease, stroke, liver cirrhosis, nephritis and other serious complications;
13. Those who have a history of psychotropic drug abuse and cannot quit or have a history of psychiatric impairment；
14. Participants with an allergic constitution, known sensitivity to human serum albumin, cyclophosphamide, fludarabine and interleukin 2;
15. Those with bleeding or thromboembolic tendency：bleeding symptoms of clinical significance or a clear tendency to bleeding within 2 weeks prior to entering the study. And those with hereditary or acquired bleeding and thrombotic tendencies； serious arterial/venous thromboembolic events occurred in the previous 6 months;
16. Other severe, acute or chronic medical or mental illnesses that in the investigator's judgement will might be increase the risk associated with the patient's participation in the study or interfere with interpretation of research results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate（ORR） | At 12months after the TCR-T cell infusion
  The objective response rate is calculated based on the patient population with measurable lesions at baseline, with efficacy determined by comparing tumor burden before and after treatment. According to RECIST 1.1 criteria，Complete Response (CR): Disappearance of all target lesions with no new lesions. Partial Response (PR): ≥30% reduction in the sum of diameters of target lesions. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions or appearance of new lesions. Stable Disease (SD): Changes not meeting any of the above thresholds.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | 1、3、7、14、28days and 2months、3 months、6 months、9 months、12months after the TCR-T cell infusion
  Peak plasma concentration (Cmax) refers to the maximum concentration of TCR-T cells in peripheral blood after the TCR-T cells infusion.
Area under the plasma concentration versus time curve (AUC) | 1、3、7、14、28days and 2months、3 months、6 months、9 months、12months after the TCR-T cell infusion
  Area under the plasma concentration versus time curve (AUC) is used to access the absorbed TCR-T cells dose into human blood circulation after TCR-T cells injection.
Peak time (Tmax) | 1、3、7、14、28days and 2months、3 months、6 months、9 months、12months after the TCR-T cell infusion
  Peak time (Tmax) refers to the time when the blood concentration reaches the peak after TCR-T cells injection.
Cell number of TCR-T cells in peripheral blood | 1、3、7、14、28days and 2months、3 months、6 months、9 months、12months after the TCR-T cell infusion
  Cell numbers of TCR-T cells after the injection of TCR-T cells
Peak value of cytokines | 1、3、7、14、28days and 2months、3 months、6 months、9 months、12months after the TCR-T cell infusion
  The peak value of cytokines within 1 month after TCR-T cell infusion .
Adverse events | 12months after TCR-T infusion
  The type, incidence and severity of adverse events include abnormal laboratory examination results with clinical significance after treatment, abnormal physical examination and blood examination results, bone marrow examination results, etc. Clinical and laboratory adverse events will be classified according to the National Cancer Institute general terminology standard for adverse events (NCI CTCAE) version 5.0.
duration of response(DOR) | 12months after TCR-T infusion
  DOR is defined as the time from the first confirmed objective response to disease progression or recurrence.
The overall survival(OS) | At 12months after the TCR-T cell infusion
  The overall survival period refers to the time of the TCR-T infusion to the death of the patient for any cause.
Progression free survival (PFS) | At 12months after the TCR-T cell infusion
  Progression free survival refers to the time from TCR-T infusion to the first occurrence of disease or death from any cause.According to RECIST version 1.1, the tumor evaluation of all subjects will be evaluated within 12 months after TCR-T treatment.
Time to progression (TTP) | 12months after the TCR-T cell infusion
  Time to progression (TTP) refers to the time from TCR-T infusion to objective tumor progression.According to RECIST version 1.1, the tumor evaluation of all subjects will be evaluated within 12 months after TCR-T treatment.
Event free survival period | At 12months after the TCR-T cell infusion
  The event free survival period (until the time of treatment failure) refers to the time from entering the trial to any treatment failure, including disease progression or cessation of treatment for any reason (such as disease progression, toxic reactions, subject willingness, initiation of new treatment without clear progression, or death).According to RECIST version 1.1, the tumor evaluation of all subjects will be evaluated within 12 months after TCR-T treatment.
The disease-free survival period | At 12months after the TCR-T cell infusion
  The disease-free survival period refers to the time from obtaining disease-free status or reaching complete response until recurrence or death due to acute toxicity of tumors or treatment.
The duration of efficacy | At 12months after the TCR-T cell infusion
  The duration of efficacy refers to the time from reaching the treatment effectiveness (i.e. CR or PR) standard until the first definite recurrence or progression is achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Zhang, MD, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Leidner R, Sanjuan Silva N, Huang H, Sprott D, Zheng C, Shih YP, Leung A, Payne R, Sutcliffe K, Cramer J, Rosenberg SA, Fox BA, Urba WJ, Tran E. Neoantigen T-Cell Receptor Gene Therapy in Pancreatic Cancer. N Engl J Med. 2022 Jun 2;386(22):2112-2119. doi: 10.1056/NEJMoa2119662. PMID 35648703
- [Background] Tran E, Robbins PF, Lu YC, Prickett TD, Gartner JJ, Jia L, Pasetto A, Zheng Z, Ray S, Groh EM, Kriley IR, Rosenberg SA. T-Cell Transfer Therapy Targeting Mutant KRAS in Cancer. N Engl J Med. 2016 Dec 8;375(23):2255-2262. doi: 10.1056/NEJMoa1609279. PMID 27959684
- [Background] Tran E, Ahmadzadeh M, Lu YC, Gros A, Turcotte S, Robbins PF, Gartner JJ, Zheng Z, Li YF, Ray S, Wunderlich JR, Somerville RP, Rosenberg SA. Immunogenicity of somatic mutations in human gastrointestinal cancers. Science. 2015 Dec 11;350(6266):1387-90. doi: 10.1126/science.aad1253. Epub 2015 Oct 29. PMID 26516200
- [Background] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403
- [Background] Morgan RA, Dudley ME, Wunderlich JR, Hughes MS, Yang JC, Sherry RM, Royal RE, Topalian SL, Kammula US, Restifo NP, Zheng Z, Nahvi A, de Vries CR, Rogers-Freezer LJ, Mavroukakis SA, Rosenberg SA. Cancer regression in patients after transfer of genetically engineered lymphocytes. Science. 2006 Oct 6;314(5796):126-9. doi: 10.1126/science.1129003. Epub 2006 Aug 31. PMID 16946036
- [Background] Morkel M, Riemer P, Blaker H, Sers C. Similar but different: distinct roles for KRAS and BRAF oncogenes in colorectal cancer development and therapy resistance. Oncotarget. 2015 Aug 28;6(25):20785-800. doi: 10.18632/oncotarget.4750. PMID 26299805
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Beatty GL, O'Hara MH, Lacey SF, Torigian DA, Nazimuddin F, Chen F, Kulikovskaya IM, Soulen MC, McGarvey M, Nelson AM, Gladney WL, Levine BL, Melenhorst JJ, Plesa G, June CH. Activity of Mesothelin-Specific Chimeric Antigen Receptor T Cells Against Pancreatic Carcinoma Metastases in a Phase 1 Trial. Gastroenterology. 2018 Jul;155(1):29-32. doi: 10.1053/j.gastro.2018.03.029. Epub 2018 Mar 20. PMID 29567081